CLINICAL TRIAL: NCT03837288
Title: Cervical Cerclage for Singleton Pregnant on Vaginal Progesterone With Progressive Cervical Length Shortening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Manal Mohammed Fawzy, Principle invistigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Trial
Record Dates: First submitted 2019-01-08; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Preterm Labor; Cervical Incompetence
Keywords: preterm labor; cerclage
MeSH Terms: conditions — Obstetric Labor, Premature; Uterine Cervical Incompetence | interventions — Cerclage, Cervical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal progesterone only (No Intervention): continue on vaginal progesterone only
- Cervical cerclage plus vaginal progesterone (Experimental): cerclage with vaginal progesterone.
  Interventions: Procedure: Cerclage

INTERVENTIONS:
Procedure: Cerclage — Cervical cerclage under effect of spinal anaesthesia
  Arms: Cervical cerclage plus vaginal progesterone

SUMMARY:
The aim of this study is to

Determine whether cerclage with vaginal progesterone will:

1. Reduce the overall spontaneous preterm birth rate.
2. Prolong pregnancy latency.
3. Improve neonatal outcome. Compared to vaginal progesterone only, in patients with progressive cervical shortening.

Research question:

Does cervical cerclage reduce the overall spontaneous preterm births in patients with progressive cervical shortening.

Research Hypothesis In this current study, the investigators hypothesize that cervical cerclage reduces spontaneous preterm births in patients with progressive cervical shortening on vaginal progesterone only.

DETAILED DESCRIPTION:
A randomized controlled trial The study will be done in Ain Shams University Hospital including women attending antenatal care clinic in Ain Shams University Hospital.

All patients entering the trial will be counselled and will sign a written consent explaining the details of the trial. All the patients included in this study will undergo routine Fetal anomaly scan at 18-24 weeks.Patients with cervical length < 20 mm in routine anomaly scan will :

1. Receive vaginal progesterone suppositories 200 mg daily.. (All patients will be continued with vaginal progesterone until 37 completed weeks or until they develop preterm rupture of membrane or preterm delivery).
2. Undergo routine follow up of cervical length every 1 to 2 weeks. Patients with progressive shortening of cervical length less than 10 mm during routine follow up, will have the option of continuing vaginal progesterone daily (Progesterone 200 mg vaginal suppositories) alone, or having cervical cerclage placed in addition to daily vaginal progesterone.

In cerclage group: all patients will sign a written consent for approval of cervical cerclage.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged: 20-38 years old.
2. Single living fetus.
3. The patient does not have history of preterm labor (before 37 weeks of gestation)
4. No history of cervical or uterine anomalies.

Exclusion Criteria:

1. Congenital anomalies in the fetus discovered during the follow up.
2. History of spontaneous preterm births.
3. Evidence of imminent delivery, or uterine contractions.
4. Evidence of rupture of membranes, or intra amniotic infection.
5. Intra uterine fetal death.
6. Uterine or cervical anomalies.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Singleton pregnant.
Enrollment: 60 (Estimated)
Dates: Start 2019-04-22 (Estimated); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-10-22 (Estimated)

PRIMARY OUTCOMES:
Gestational age of delivery | <37 weeks
  After 37 weeks of pregnancy

SECONDARY OUTCOMES:
New born birth weight | At time of birth
  less than 2 kg

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Shahawy, Study Director — Ain Shams University
Locations (1):
- AinshamsU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eleje GU, Eke AC, Ikechebelu JI, Ezebialu IU, Okam PC, Ilika CP. Cervical stitch (cerclage) in combination with other treatments for preventing spontaneous preterm birth in singleton pregnancies. Cochrane Database Syst Rev. 2020 Sep 24;9(9):CD012871. doi: 10.1002/14651858.CD012871.pub2. PMID 32970845